CLINICAL TRIAL: NCT02079545
Title: A Phase 1, Randomized, Open-label, Parallel-design Study to Assess Absolute Bioavailability and Single-dose Pharmacokinetics Following Subcutaneous Administration of Sirukumab Delivered By A Pre-filled Syringe Fitted With UltraSafe Passive™ Delivery System or an Autoinjector in Healthy Male Subjects
Brief Title: Bioavailability and Pharmacokinetics Study of Sirukumab in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CR103367; CNTO136NAP1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-03-04; First posted 2014-03-05 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Healthy; Bioavailability; Pharmacokinetics; Sirukumab; Subcutaneous; Male
MeSH Terms: interventions — sirukumab; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): 18 participants will receive a single intravenous (IV) infusion of 100 mg sirukumab
  Interventions: Drug: Sirukumab (IV infusion)
- Group 2 (Experimental): 18 participants will receive a single subcutaneous (SC) injection of 50 mg sirukumab using a Pre-filled Syringe (PFS) fitted with the UltraSafe Passive™ Delivery System (PFS-U)
  Interventions: Drug: Sirukumab (SC injection with PFS-U)
- Group 3 (Experimental): 18 participants will receive a single SC injection of 50 mg sirukumab using the SmartJect™ Autoinjector (PFS-AI)
  Interventions: Drug: Sirukumab (SC injection with PFS-AI)
- Group 4 (Experimental): 42 participants will receive a single SC injection of 100 mg sirukumab using a PFS-U
  Interventions: Drug: Sirukumab (SC injection with PFS-U)
- Group 5 (Experimental): 42 participants will receive a single SC injection of 100 mg sirukumab using a PFS-AI
  Interventions: Drug: Sirukumab (SC injection with PFS-AI)

INTERVENTIONS:
Drug: Sirukumab (IV infusion) — Participants will receive a single IV infusion of 100 mg sirukumab.
  Arms: Group 1
Drug: Sirukumab (SC injection with PFS-U) — Participants will receive a single SC injection of 50 mg sirukumab with PFS-U.
  Arms: Group 2
Drug: Sirukumab (SC injection with PFS-AI) — Participants will receive a single SC injection of 50 mg sirukumab with PFS-AI.
  Arms: Group 3
Drug: Sirukumab (SC injection with PFS-U) — Participants will receive a single SC injection of 100 mg sirukumab with PFS-U.
  Arms: Group 4
Drug: Sirukumab (SC injection with PFS-AI) — Participants will receive a single SC injection of 100 mg sirukumab with PFS-AI.
  Arms: Group 5

SUMMARY:
The purpose of the study is to assess the bioavailability (the extent to which a medication becomes available to the body) of subcutaneously (under the skin using a needle) administered sirukumab and to compare the pharmacokinetics of sirukumab administered subcutaneously using a pre-filled syringe fitted with the UltraSafe Passive™ Delivery system (PFS-U) with the SmartJect™ Autoinjector (PFS-AI) in healthy male participants.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention), parallel-group (each group of participants will be treated at the same time), multicenter; single-dose study. Approximately 138 participants will be randomly allocated in a 3:3:3:7:7 ratio to 1 of the 5 treatment groups as follows: Group 1 (a single intravenous infusion of 100 mg sirukumab), Group 2 (a single subcutaneous [SC] injection of 50 mg sirukumab with PFS-U), Group 3 (a single SC injection of 50 mg sirukumab with PFS-AI, Group 4 (a single SC injection of 100 mg sirukumab with PFS-U), and Group 5 (a single SC injection of 100 mg sirukumab with PFS-AI). Randomization will be stratified by body weight (50.0 kg to <70.0 kg, 70.0 kg to <85.0 kg, 85.0 kg to 100.0 kg). Participants will be hospitalized in the study unit for administration of study drug and will be discharged after completion of all scheduled assessments on Day 5. Participants will be required to return to the study unit for outpatient visits on Days 6 and 7, followed by weekly/biweekly outpatient visits, and then a safety follow-up for a total of 13 weeks after study drug administration. Safety evaluations will include assessment of adverse events, physical examination, vital signs, injection site and infusion reactions, electrocardiogram, and clinical laboratory tests. The maximum study duration for each participant will be 120 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have a weight in the range of 50.0 kg to 100.0 kg, inclusive
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram performed at screening
* Each participant must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study
* Must be willing and able to adhere to the study visit schedule and other protocol requirements
* Must agree to abstain from alcohol intake 48 hours before administration of study agent and during the inpatient period of the study

Exclusion Criteria:

* Have any known malignancy or history of malignancy, except for nonmelanoma skin cancer that has been treated with no evidence of recurrence for at least 3 months before Day 1
* Have a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly
* Have any underlying physical or psychological medical condition that, in the opinion of the investigator, would make it unlikely that the participant will complete the study
* Have evidence of any chronic medical condition requiring prescription medications (eg, hypertension, elevated cholesterol/triglycerides, asthma, or diabetes)
* Have a history of or current elevations in triglycerides that required treatment

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of 100 mg sirukumab administered subcutanoeusly | Up to Week 13
  Bioavailability will be evaluated by using the formula: AUC from time zero to infinity with extrapolation of the terminal phase of SC injection divided by AUC from time zero to infinity with extrapolation of the terminal phase of IV infusion of sirukumab and multiplied by 100.
Maximum Observed Serum Concentration (Cmax) of 100 mg sirukumab administered subcutanoeusly | Up to Week 13
  The Serum Concentration (Cmax) is defined as maximum observed analyte concentration.
Area Under the Serum Concentration-Time Curve From Time Zero to 77 days (AUC0-77d) of 100 mg sirukumab administered subcutanoeusly | Up to Week 13

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to Week 13
Immunogenicity of sirukumab | Up to Week 13
  Serum levels of antibodies to sirukumab will be used to evaluate potential immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Tempe, Arizona
  - Lincoln, Nebraska